CLINICAL TRIAL: NCT01807611
Title: Haploidentical Donor Hematopoietic Progenitor Cell and Natural Killer Cell Transplantation With a TLI Based Conditioning Regimen in Patients With Hematologic Malignancies
Brief Title: Haploidentical Donor Hematopoietic Progenitor Cell and NK Cell Transplantation for Hematologic Malignancy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Assisi Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAPNK1; NCI-2013-00609 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2013-03-05; First posted 2013-03-08 (Estimated); Results first posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-08

CONDITIONS: Leukemia; Lymphoma
Keywords: Haploidentical donor transplantation; NK cell
MeSH Terms: conditions — Leukemia; Lymphoma | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Thiotepa; Melphalan; Granulocyte Colony-Stimulating Factor; Filgrastim; Mesna; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Transplant Recipients (Experimental): Participants undergo a preparative regimen of total lymphoid irradiation, fludarabine, cyclophosphamide, fludarabine, thiotepa, melphalan, and mycophenolate mofetil, followed by HPC,A infusion and TC-NK infusion. They also receive G-CSF and mesna.
  Cells for infusion are prepared using the CliniMACS System.
  Interventions: Radiation: Total Lymphoid Irradiation; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Thiotepa; Drug: Melphalan; Biological: HPC,A Infusion; Biological: TC-NK Infusion; Biological: G-CSF; Drug: Mesna; Device: CliniMACS; Drug: Mycophenolate mofetil

INTERVENTIONS:
Radiation: Total Lymphoid Irradiation — Participants receive total lymphoid irradiation over four doses.
  Other Names: TLI
Drug: Fludarabine — Given IV.
  Other Names: Fludara
Drug: Cyclophosphamide — Given IV.
  Other Names: Cytoxan
Drug: Thiotepa — Given IV.
  Other Names: Thioplex(R) by Immunex; TESPA; TSPA
Drug: Melphalan — Given IV.
  Other Names: L-phenylalanine mustard; Phenylalanine Mustard; L-PAM; L-sarcolysin; Alkeran(R)
Biological: HPC,A Infusion — Participants received infusions of HPC,A (CD34+ selected) and HPC,A (CD45RA depleted).
Biological: TC-NK Infusion — Participants receive infusions of TC-NK.
Biological: G-CSF — Participants receive G-CSF subcutaneously or intravenously.
  Donors receive G-CSF subcutaneously during cell mobilization.
  Other Names: Granulocyte Colony-Stimulating Factor; Filgrastim; Neupogen(R)
Drug: Mesna — Mesna is generally dosed at approximately 25% of the cyclophosphamide dose. It is generally given intravenously prior to and again at 3, 6 and 9 hours following each dose of cyclophosphamide.
  Other Names: Mesnex
Device: CliniMACS — The mechanism of action of the CliniMACS Cell Selection System is based on magnetic-activated cell sorting (MACS). The CliniMACS device is a powerful tool for the isolation of many cell types from heterogeneous cell mixtures, (e.g. apheresis products). These can then be separated in a magnetic field using an immunomagnetic label specific for the cell type of interest, such as CD3+ human T cells.
  Other Names: Cell Selection System
Drug: Mycophenolate mofetil — Given intravenously or orally.
  Other Names: MMF; CellCept®

SUMMARY:
In this study, participants with high-risk hematologic malignancies undergoing hematopoietic cell transplantation (HCT), who do not have a suitable human leukocyte antigen (HLA) matched related/sibling donor (MSD) or matched unrelated donor (MUD) identified, will receive a haploidentical donor HCT with additional natural killer (NK) cells.

The investigators anticipate enrollment of 75 donors and 75 recipients.

PRIMARY OBJECTIVE:

* To estimate the rate of successful engraftment at day +42 post-transplant in patients who receive haploidentical donor stem cell plus NK cell transplantation with TLI based conditioning regimen for high risk hematologic malignancy.

SECONDARY OBJECTIVES:

* Estimate the incidence of malignant relapse, event-free survival, and overall survival at one-year post-transplantation.
* Estimate incidence and severity of acute and chronic (GVHD).
* Estimate the rate of transplant related mortality (TRM) in the first 100 days after transplantation.

DETAILED DESCRIPTION:
Donors will undergo G-CSF mobilization of peripheral blood stem cells (PBSC) prior to undergoing two apheresis collections of hematopoietic progenitor cells (HPC,A) and one apheresis collection of therapeutic cell product of purified natural killer cells (TC-NK).

The HPC products will be T-cell depleted (TCD) using the investigational CliniMACS device. CD34+ enrichment and CD45RA depletion will be utilized on sequential HPC grafts.

Participants will undergo a preparative regimen of total lymphoid irradiation, fludarabine, cyclophosphamide, granulocyte colony stimulating factor (G-CSF), thiotepa, and melphalan. This is followed by infusions of donor cells that have been prepared using the CliniMACS system: HPC,A (CD34+ selected), HPC,A (CD45RA depleted), and TC-NK.

ELIGIBILITY:
Inclusion Criteria - Transplant Recipients:

* Age less than or equal to 21 years.
* Does not have a suitable MSD or volunteer MUD available in the necessary time for stem cell donation.
* Has a suitable single haplotype matched (≥ 3 of 6) and family member donor.
* High risk hematologic malignancy.
* If prior CNS leukemia, it must be treated and in CNS CR
* Does not have any other active malignancy other than the one for which this HCT is indicated.
* No prior allogeneic HCT, and no autologous HCT within the previous 12 months.
* Patient must fulfill pre-transplant evaluation

Inclusion Criteria - Haploidentical Donor:

* At least single haplotype matched (≥ 3 of 6) family member
* At least 18 years of age.
* HIV negative.
* Not pregnant as confirmed by negative serum or urine pregnancy test within 14 days prior to enrollment (if female).
* Not breast feeding.
* Regarding eligibility, is identified as either: (1) Completed the process of donor eligibility determination as outlined in 21 CFR 1271 and agency guidance; OR (2) Does not meet 21 CFR 1271 eligibility requirements, but has a declaration of urgent medical need completed by the principal investigator or physician sub-investigator per 21 CFR 1271.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2013-05-16 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon M. Triplett, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Naik S, Li Y, Talleur AC, Selukar S, Ashcraft E, Cheng C, Madden RM, Mamcarz E, Qudeimat A, Sharma A, Srinivasan A, Suliman AY, Epperly R, Obeng EA, Velasquez MP, Langfitt D, Schell S, Metais JY, Arnold PY, Hijano DR, Maron G, Merchant TE, Akel S, Leung W, Gottschalk S, Triplett BM. Memory T-cell enriched haploidentical transplantation with NK cell addback results in promising long-term outcomes: a phase II trial. J Hematol Oncol. 2024 Jun 27;17(1):50. doi: 10.1186/s13045-024-01567-0. PMID 38937803
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There are in total 82 transplant recipients enrolled.
Groups:
- Transplant Recipients: Participants undergo a preparative regimen of total lymphoid irradiation, fludarabine, cyclophosphamide, fludarabine, thiotepa, melphalan, and mycophenolate mofetil, followed by HPC,A infusion and TC-NK infusion. They also receive G-CSF and mesna.
  Cells for infusion are prepared using the CliniMACS System. Total Lymphoid Irradiation: Participants receive total lymphoid irradiation over four doses. Fludarabine: Given IV.
  Cyclophosphamide: Given IV. Thiotepa: Given IV. Melphalan: Given IV. HPC,A Infusion: Participants received infusions of HPC,A (CD34+ selected) and HPC,A (CD45RA depleted). TC-NK Infusion: Participants receive infusions of TC-NK.
  G-CSF: Participants receive G-CSF subcutaneously or intravenously. Donors receive G-CSF subcutaneously during cell mobilization.
  Mesna: Mesna is generally dosed at approximately 25% of the cyclophosphamide dose. It is generally given intravenously prior to and again at 3, 6 and 9 hours following each dose of cyclophosphamide.
  CliniMACS: The mechanism of action of the CliniMACS Cell Selection System is based on magnetic-activated cell sorting (MACS). The CliniMACS device is a powerful tool for the isolation of many cell types from heterogeneous cell mixtures, (e.g. apheresis products). These can then be separated in a magnetic field using an immunomagnetic label specific for the cell type of interest, such as CD3+ human T cells.
  Mycophenolate mofetil: Given intravenously or orally.
Period: Overall Study
Arm/Group | Transplant Recipients
Started | 82
Completed | 78
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Age was evaluated at the time of transplantation.
Groups:
- Experimental: Transplant Recipients: Participants meeting eligibility criteria and who completed study therapy: haploidentical stem cell transplantation with additional natural killer (NK) cells and total lymphoid irradiation (TLI) based conditioning regimen. Participants who received a therapeutic variance (maraviroc) are excluded.
Arm/Group | Experimental: Transplant Recipients
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 63
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.5 (6.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 52
  More than one race | 3
  Unknown or Not Reported | 0
Donor relationship to patient: Father, Mother, Sibling, Other. [Count of Participants; unit: Participants]
  Father | 35
  Mother | 31
  Sibling | 4
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Transplant Recipients With Successful Engraftment
Description: Neutrophil engraftment will be determined using the parameters put forth by the Center for International Blood and Marrow Registry. Assessments will be made upon review of daily complete blood count and serial chimerism studies. Successful engraftment for the purposes of this objective will be patients who do not experience graft failure.
Time Frame: 42 days post engraftment
Population: Participants meeting eligibility criteria and who completed study therapy: haploidentical stem cell transplantation with additional natural killer (NK) cells and total lymphoid irradiation (TLI) based conditioning regimen. Participants who received a therapeutic variance (maraviroc) are excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Transplant Recipients
Number analyzed (Participants) | 72
Participants | 70

2. Secondary Outcome: Number of Transplant Recipients With Malignant Relapse
Description: Bone marrow studies for disease status evaluation will be performed at 1-year post-transplant. Testing will include a research evaluation for minimal residual disease.
Time Frame: One-year post-transplantation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Transplant Recipients
Number analyzed (Participants) | 72
Participants | 18

3. Secondary Outcome: Event-free Survival
Description: The one-year event free survival is defined by the patient who has neither experienced relapse nor death within one year after post transplantation. And the rate is calculated by computing the ratio between total number of one year event free survival patients and the total number of patients.
Time Frame: One year post-transplantation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Transplant Recipients
Number analyzed (Participants) | 72
Participants | 49

4. Secondary Outcome: Overall Survival
Description: The one-year survival is defined by the patient who has not died within one year after post transplantation. And the rate is calculated by computing the ratio between total number of one year survival patients and the total number of patients.
Time Frame: one year post-transplantation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Transplant Recipients
Number analyzed (Participants) | 72
Participants | 59

5. Secondary Outcome: Number of Transplant Recipients With Acute and/or Chronic Graft Versus Host Disease (GVHD)
Description: Acute and chronic graft-vs.-host disease will be evaluated using the standard grading criteria. The estimate will be the number of recipients who experienced GVHD divided by the total number of patients considered in this group.
Time Frame: 100 days post-transplant for acute GVHD; one year post-transplant for chronic GVHD .
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Number of Transplant Recipients With Acute Graft Versus Host Disease (aGVHD); Number of Transplant Recipients With Chronic Graft Versus Host Disease (cGVHD): Participants meeting eligibility criteria and who completed study therapy: haploidentical stem cell transplantation with additional natural killer (NK) cells and total lymphoid irradiation (TLI) based conditioning regimen. Participants who received a therapeutic variance (maraviroc) are excluded.
Arm/Group | Number of Transplant Recipients With Acute Graft Versus Host Disease (aGVHD) | Number of Transplant Recipients With Chronic Graft Versus Host Disease (cGVHD)
Number analyzed (Participants) | 72 | 72
Participants | 24 | 16

6. Secondary Outcome: Number of Transplant Recipients With Transplant-related Mortality (TRM)
Description: Estimate the proportion of patients died within 100 days after the transplantation who has not experienced a relapse. The estimate will be the number of TRM divides the total number of patients considered in this group.
Time Frame: In the first 100 days after transplantation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Transplant Recipients
Number analyzed (Participants) | 72
Participants | 4

7. Secondary Outcome: Severity of Acute Graft Versus Host Disease (aGVHD)
Description: Ongoing assessment of toxicity will be done using the NCI CTCAE version 3.0. Acute and chronic graft-vs.-host disease will be evaluated using the standard grading criteria. The severity of acute GvHD and chronic GvHD will be described. The analysis for this objective will be performed when the last evaluable participant has been followed for 100 days post transplant. Acute GvHD is graded from 1-4 with 4 being the worst outcome.
Time Frame: 100 days post-transplant for acute GVHD.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Severity of Acute Graft Versus Host Disease (aGVHD): Ongoing assessment of toxicity will be done using the NCI CTCAE version 3.0. Acute and chronic graft-vs.-host disease will be evaluated using the standard grading criteria. The severity of acute GvHD and chronic GvHD will be described. The analysis for this objective will be performed when the last evaluable participant has been followed for 100 days post-transplant.
Arm/Group | Severity of Acute Graft Versus Host Disease (aGVHD)
Number analyzed (Participants) | 72
Participants
  No aGVHD within 100 days | 48
  Grade 1 aGVHD within 100 days | 2
  Grade 2 aGVHD within 100 days | 2
  Grade 3 aGVHD within 100 days | 16
  Grade 4 aGVHD within 100 days | 4

8. Secondary Outcome: Severity of Chronic Graft Versus Host Disease (cGVHD)
Description: Ongoing assessment of toxicity will be done using the NCI CTCAE version 3.0. Acute and chronic graft-vs.-host disease will be evaluated using the standard grading criteria. The severity of acute GvHD and chronic GvHD will be described. The analysis for this objective will be performed when the last evaluable participant has been followed for 1 year post-transplant. Chronic GvHD is graded as "mild", "moderate" or "severe" with "severe" being the worst outcome.
Time Frame: 1 year post-transplant for chronic GVHD .
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Severity of Chronic Graft Versus Host Disease (cGVHD): Ongoing assessment of toxicity will be done using the NCI CTCAE version 3.0. Acute and chronic graft-vs.-host disease will be evaluated using the standard grading criteria. The severity of acute GvHD and chronic GvHD will be described. The analysis for this objective will be performed when the last evaluable participant has been followed for 1 year post-transplant. Chronic GvHD is graded as "mild", "moderate" or "severe" with "severe" being the worst outcome.
Arm/Group | Severity of Chronic Graft Versus Host Disease (cGVHD)
Number analyzed (Participants) | 72
Participants
  No cGVHD within 1st year | 56
  Mild | 6
  Moderate | 5
  Severe | 5

ADVERSE EVENTS:
Time Frame: Transplant recipients will be followed for adverse events from the start of conditioning and throughout the first-year post-transplant
Description: Recipient participants were followed for all NCI Grade III-V adverse events from the start of conditioning through the first-year post HCT, regardless of their relationship to the treatment given. Clinically significant NCI Grade I-II adverse events that are judged to be related/possibly related may be collected per the discretion and judgment of the PI. Adverse events that affected more than 5 participants are included in this description.
Groups:
- Experimental: Transplant Recipients: Participants meeting eligibility criteria and who completed study therapy: haploidentical stem cell transplantation with additional natural killer (NK) cells and total lymphoid irradiation (TLI) based conditioning regimen. Participants who received a therapeutic variance (maraviroc) are included.
Arm/Group | Experimental: Transplant Recipients
All-Cause Mortality (participants affected / at risk) | 14/78
Serious Adverse Events (participants affected / at risk) | 56/78
Other Adverse Events (participants affected / at risk) | 78/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Transplant Recipients (N=78)
Febrile Without Neutropenia (Infections and infestations) | 17
Febrile Neutropenia (Infections and infestations) | 10
Pericardial Effusion (Cardiac disorders) | 7
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 7
Hypotension (Cardiac disorders) | 6
Acute Kidney Injury (Renal and urinary disorders) | 5
Infection, Staphylococcus Epidermidis, Blood (Infections and infestations) | 5
Seizure (Nervous system disorders) | 5
Fever (General disorders) | 4
Hemorrhage, Pulmonary (Blood and lymphatic system disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Transplant Recipients (N=78)
Febrile Neutropenia (Infections and infestations) | 67
Mucositis (Gastrointestinal disorders) | 50
Infection, Clostridium Difficile, Stool (Infections and infestations) | 33
Infection, Human Herpesvirus 6, Blood (Infections and infestations) | 32
Febrile Without Neutropenia (Infections and infestations) | 28
Infection, Adenovirus, Stool (Infections and infestations) | 26
Engraftment Syndrome (Immune system disorders) | 24
Infection, Candida, Oral (Infections and infestations) | 22
Hypertension (Cardiac disorders) | 20
Infection, Cytomegalovirus, Blood (Infections and infestations) | 18
Tachycardia (finding) (Cardiac disorders) | 16
Nausea (Gastrointestinal disorders) | 15
Infection, BK Virus, Urine (Infections and infestations) | 12
Diarrhea (Gastrointestinal disorders) | 11
Hemorrhagic Cystitis (Renal and urinary disorders) | 11
Hypotension (Cardiac disorders) | 10
Infection, Rotavirus, Stool (Infections and infestations) | 10
Cytokine Release Syndrome (Immune system disorders) | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8
Acute Kidney Injury (Renal and urinary disorders) | 7
Infection, Staphylococcus Epidermidis, Blood (Infections and infestations) | 7
Alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase) (SGPT) level abnormal (finding) (Metabolism and nutrition disorders) | 6
Diastolic dysfunction (finding) (Cardiac disorders) | 6
Infection, Adenovirus, Blood (Infections and infestations) | 6
Infection, Epstein Barr Virus, Blood (Infections and infestations) | 6
Infection, Adenovirus, Respiratory Tract (Infections and infestations) | 5
Infection, Norovirus, Stool (Infections and infestations) | 5
Transaminitis (Metabolism and nutrition disorders) | 5
Confusion (Nervous system disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 4
Epistaxis (Blood and lymphatic system disorders) | 4
Infection, BK Virus, Blood (Infections and infestations) | 4
Infection, Streptococcus Viridans, Blood (Infections and infestations) | 4
Pneumatosis Intestinalis (Gastrointestinal disorders) | 4
Weight Loss (Metabolism and nutrition disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT01807611/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT01807611/ICF_001.pdf